CLINICAL TRIAL: NCT05847062
Title: Clinical Study to Analyze the Functional, Radiological, and Strength Results in Lateralized Models and Inverted Arthroplasty Medializations
Brief Title: Clinical Trial to Analyze Lateralized Models and Medializations of Inverted Arthroplasty.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yaiza Lopiz Morales (Other)
Responsible Party: Sponsor-Investigator, Yaiza Lopiz Morales, Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22/016-EC_X
Record Dates: First submitted 2023-02-28; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Rotator Cuff Arthropathy; Glenohumeral Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This is an experimental, prospective, unblinded, randomized, comparative clinical trial between patients carrying two types of prosthetic implants with a different biomechanical design based on medialization or lateralization of the center of rotation of the inverted prosthesis.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients will be randomized to assign them to one or another study group, which will be carried out by an independent assistant, who will generate a random sequence that will be unknown to the investigators. Each patient will be given a sealed and numbered envelope to choose from, in which the randomized group in which he/she has been included will be determined. The study will be blinded for the patient and rehabilitator but not for the surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients operated on by means of an inverted shoulder prosthesis with medialized component (Active Comparator): patients meeting the inclusion criteria who underwent surgery for a rotator cuff tear using an inverted shoulder prosthesis with a medially rotated center of rotation.
  Interventions: Procedure: reverse shoulder arthroplasty
- patients operated by means of inverted shoulder prosthesis with lateralized component (Active Comparator): patients meeting the inclusion criteria who underwent surgery for a rotator cuff tear using an inverted shoulder prosthesis with a lateralized center of rotation.
  Interventions: Procedure: reverse shoulder arthroplasty

INTERVENTIONS:
Procedure: reverse shoulder arthroplasty — The patient will be admitted to undergo reconstructive surgery of the arthropathy, by means of one of the two mentioned Inverted Arthroplasty implants. The patient will be operated following always the same surgical technique with the same protocol (position, anesthesia, antibiotic prophylaxis...) and by one of the three surgeons of the shoulder unit, being always at least two of them present in each of the interventions. Both the implants used and the complications occurring during surgery or in the immediate postoperative period will be recorded.

SUMMARY:
To determine the functional outcomes, complications and muscle performance by isokinetic study of two reverse arthroplasty systems (one with medialized center of rotation and the other with lateralized center of rotation) in the treatment of rotator cuff arthropathies or irreparable cuff tears.

DETAILED DESCRIPTION:
This is an experimental, prospective, unblinded, randomized, comparative clinical trial between patients with two types of prosthetic implants (inverted arthroplasty with medialized center of rotation vs inverted arthroplasty with lateralized center of rotation). Those male or female patients who meet the inclusion criteria will be selected to form part of one of the two randomly distributed study groups. Sample size Based on studies with similar characteristics but where lateralization is not performed with the implant but with a bone graft would require a sample size of 34 patients (17 in each group) assuming 20% losses with a Type I error of 0. 05 and a statistical power of 80% to show a difference of 10 points on the Constant scale (the minimal clinically important difference on the Constant scale for reverse arthroplasty is described as 8 points in previous comparative studies so we consider the detection of a difference of 10 to be sufficient. The minimal clinically important difference for function and strength in patients undergoing reverse shoulder arthroplasty. The final N needed would be 42 patients (21 per group). A randomization of patients will be performed to assign them to one or the other study group, which will be carried out by an independent assistant, who will generate a random sequence that will be unknown to the investigators. Each patient will be given a sealed and numbered envelope to choose from, in which the randomized group in which he/she has been included will be determined. The study will be blinded for the patient and rehabilitator but not for the surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over 65 years of age with rotator cuff arthropathy refractory to conservative treatment after six months.
2. Ability to understand the information sheet, informed consent and evaluation scales.

   Exclusion Criteria:

   Patients with sequelae of fractures, rheumatoid arthritis, avascular necrosis, primary glenohumeral arthrosis, revision surgeries that have required conversion to a ATHI
3. Patients in whom another surgical procedure has been associated with ATHI such as a tendon transfer
4. Glenoid bone defects in the horizontal plane (Type B2 and C of the Walch classification) or in the vertical plane (E3 Sirveaux).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
to compare functional outcomes in patients with cuff arthropathies treated with medialized ATHI or lateralized ATHI. | 24 Months
  To compare functional outcomes (Constant scale score) 24 months after surgery in patients over 65 years of age with cuff arthropathies treated with either of two options: Medialized ATHI or lateralized ATHI. the score ranges from 0-100 points. The higher the score the better the functional result

SECONDARY OUTCOMES:
Comparison of the results of the visual analog pain scale (VAS) | 24 Months
  Comparison of the results obtained in the other functional assessment scale: the visual analog pain scale (VAS).(0-10). The higher the score, the more painful
Comparison of Joint Range of Motion between the two prosthetic systems under study. | 24 Months
  Comparison of the joint range of motion (joint balance in degrees in abduction, external and internal rotation, anteversion) between the two prosthetic systems under study.
Analysis and comparison of the Maximum recorded muscle force. | 24 Months
  Maximum muscle force at any time during a repetition. Indicative of muscle force capacity (N-M, newtons per meter).
Determination and comparison of the prevalence of complications with each of the prosthetic systems. | 24 Months
  Determination and comparison of the prevalence of complications with each of the prosthetic systems used, including radiographic evaluation.
Comparison of the results of the Quick Disabilities of arm, shoulder and hand (Quick-DASH) score. | 24 Months
  Comparison of the results obtained in the other functional assessment scale: Quick Disabilities of arm, shoulder and hand (Quick-DASH) score. The score ranges from 0 to 100.
  The higher the score, the greater shoulder disability
Comparison of the results of the American Shoulder and Elbow Surgeons score | 24 Months
  Comparison of the results obtained in the other functional assessment scales: American Shoulder and Elbow Surgeons score. the the score ranges from 0 to 100, where 0 indicates a worse shoulder condition and 100 indicates best shoulder condition, so the greater the score, the lower the level of shoulder disability
Analysis and comparison of the Maximum strength as a function of weight | 24 Months
  Maximum strength as a function of weight: percentage of muscle strength recorded and normalized by body weight and compared to the set goal ( %).
Analysis and comparison of the Total work per repetition | 24 Months
  Total work per repetition: total muscle force for the repetition with the greatest amount of work. Work is indicative of the muscle's ability to produce force throughout the range of motion (measured in Joules (J)).
Analysis and comparison of the isokinetic parameter (Coefficient of variation ) | 24 Months
  Coefficient of variation : Statistical representation of the validity of the test based on the reproducibility of the exercise. Low values show higher reproducibility (%).
Analysis and comparison of the isokinetic parameters (Average power) | 24 Months
  Average power: total work divided by time. Power represents how fast a muscle can produce force (W, watts).
Analysis and comparison of the Acceleration rate | 24 Months
  Acceleration rate: total time to reach the Isokinetic speed. Indicative of the neuromuscular capacity to move the limb at the beginning of the Range of Motion (msec. milliseconds).
Analysis and comparison of the Deceleration speed | 24 Months
  Deceleration speed: total time to go from Isokinetic speed to zero speed. Indicative of the neuromuscular capacity to control the limb eccentrically at the end of the Range of Motion (msec, milliseconds).
Analysis and comparison of the isokinetic parameters (Agonist/antagonist ratio) | 24 Months
  Agonist/antagonist ratio: The ratio of the reciprocal muscle group. Excessive imbalances may predispose to joint injury.%

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos de Madrid, Madrid, Spain

REFERENCES:
- [Background] Lopiz Y, Garcia-Fernandez C, Arriaza A, Rizo B, Marcelo H, Marco F. Midterm outcomes of bone grafting in glenoid defects treated with reverse shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Sep;26(9):1581-1588. doi: 10.1016/j.jse.2017.01.017. Epub 2017 Apr 10. PMID 28408254
- [Background] Lopiz Y, Rodriguez-Gonzalez A, Martin-Albarran S, Marcelo H, Garcia-Fernandez C, Marco F. Injury to the axillary and suprascapular nerves in rotator cuff arthropathy and after reverse shoulder arthroplasty: a prospective electromyographic analysis. J Shoulder Elbow Surg. 2018 Jul;27(7):1275-1282. doi: 10.1016/j.jse.2017.12.030. Epub 2018 Feb 21. PMID 29475786
- [Background] Garcia-Fernandez C, Lopiz Y, Rizo B, Serrano-Mateo L, Alcobia-Diaz B, Rodriguez-Gonzalez A, Marco F. Reverse total shoulder arhroplasty for the treatment of failed fixation in proximal humeral fractures. Injury. 2018 Sep;49 Suppl 2:S22-S26. doi: 10.1016/j.injury.2018.06.042. PMID 30219143
- [Background] Lopiz Y, Alcobia-Diaz B, Galan-Olleros M, Garcia-Fernandez C, Picado AL, Marco F. Reverse shoulder arthroplasty versus nonoperative treatment for 3- or 4-part proximal humeral fractures in elderly patients: a prospective randomized controlled trial. J Shoulder Elbow Surg. 2019 Dec;28(12):2259-2271. doi: 10.1016/j.jse.2019.06.024. Epub 2019 Sep 6. PMID 31500986
- [Background] Lopiz Y, Garcia-Fernandez C, Vallejo-Carrasco M, Garriguez-Perez D, Achaerandio L, Tesoro-Gonzalo C, Marco F. Reverse shoulder arthroplasty for proximal humeral fracture in the elderly. Cemented or uncemented stem? Int Orthop. 2022 Mar;46(3):635-644. doi: 10.1007/s00264-021-05284-y. Epub 2022 Jan 16. PMID 35034145

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT05847062/Prot_SAP_ICF_000.pdf